CLINICAL TRIAL: NCT03979079
Title: Modeling Clinical Failure in Prostate Cancer Patients Based on a Two-stage Statistical Model
Acronym: PREDYC
Status: Completed | Type: Observational
Sponsor: Institut Bergonié (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: IB2010-PREDYC
Record Dates: First submitted 2019-06-04; First posted 2019-06-07 (Actual); Results first posted 2020-12-21 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2020-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: external beam radiation therapy

SUMMARY:
Biomarker series can indicate disease progression and predict clinical endpoints. When a treatment is prescribed depending on the biomarker, confounding by indication might be introduced if the treatment modifies the marker profile and risk of failure.

The two-stage model fitted within a Bayesian Markov Chain Monte Carlo framework is particularly flexible to account for such data. Prostate-specific antigens in prostate cancer patients treated with external beam radiation therapy can be monitored. In the presence of rising prostate-specific antigens after external beam radiation therapy, salvage hormone therapy can be prescribed to reduce both the prostate-specific antigens concentration and the risk of clinical failure, an illustration of confounding by indication. The prognostic value of hormone therapy and prostate-specific antigens trajectory on the risk of failure based on a two-stage model within a Bayesian framework to assess the role of the prostate-specific antigens profile on clinical failure while accounting for a secondary treatment prescribed by indication. the aim of this research is to model prostate specific antigens using a hierarchical piecewise linear trajectory with a random changepoint. Residual prostate-specific antigens variability can be expressed as a function of prostate-specific antigens concentration. Covariates in the survival model can include : hormone therapy, baseline characteristics, and individual predictions of the prostate-specific antigens nadir and timing and prostate-specific antigens slopes before and after the nadir as provided by the longitudinal process.

DETAILED DESCRIPTION:
The two-stage modeling approach allows estimation of the regression coefficients in a time-dependent Cox model, while addressing the limitations with the knowledge of the true marker trajectory. In the first stage, the longitudinal process is modeled using a repeated measures component model, such as a random effects model. In the second stage, estimated characteristics of the longitudinal marker trajectory, such as slopes, are included as covariates in a survival model to assess their prognostic value.

Our aim was to highlight the flexibility of a two-stage model fitted within a Bayesian Markov Chain Monte Carlo (MCMC) framework. We applied this model to assess the prognostic value of the prostate-specific antigens (PSA) profile (level and timing of the nadir; pre- and post-nadir slopes) as well as salvage hormonal treatment (HT) on the risk of clinical failure following external beam radiation therapy (EBRT) in the presence of confounding by indication. We first present the longitudinal hierarchical PSA model that we developed earlier. This model was particularly flexible since it allowed us to account for the presence of a random changepoint as well as the modeling of the residual variability as a function of the PSA concentration. We next extend the longitudinal model to a two-stage model by using estimated parameters of the longitudinal process as covariates in a Cox proportional hazards model to assess prognostic factors of clinical failure including baseline characteristics, PSA trajectory, and HT.

ELIGIBILITY:
Inclusion Criteria:

* clinically localized prostate cancer
* Clinical stage T1 to T4
* Node and metastasis negative
* Treated with external beam radiation therapy (RT).

Exclusion Criteria:

* Patients with baseline or planned hormonotherapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Dataset of 2384 men included in three cohorts: University of Michigan, Ann Arbor, MI, USA (UM); Radiation Therapy Oncology Group (RTOG 9406); and William Beaumont Hospital, Detroit, MI, USA.
Sampling Method: Non-Probability Sample
Enrollment: 2384 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carine Bellera, PhD, Principal Investigator — Institut Bergonié
Locations (1):
- INSERM, Bordeaux, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Bellera C, Proust-Lima C, Joseph L, Richaud P, Taylor J, Sandler H, Hanley J, Mathoulin-Pelissier S. A two-stage model in a Bayesian framework to estimate a survival endpoint in the presence of confounding by indication. Stat Methods Med Res. 2018 Apr;27(4):1271-1281. doi: 10.1177/0962280216660127. Epub 2016 Sep 1. PMID 27587597

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients: Eligible Prostate Cancer Patients Undergoing EBRT Treatment
Period: Overall Study
Arm/Group | Patients
Started | 2384
Completed | 2384
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Eligible Patients: Eligible Prostate Cancer Patients Undergoing EBRT Treatment
Arm/Group | Eligible Patients
Number analyzed (Participants) | 2384
Age, Continuous [Mean (Standard Deviation); unit: years] | 72 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2384
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Failure After Initiation of Radiotherapy
Description: Clinical failure is defined as any of the following events following initiation of radiotherapy: distant metastases, nodal recurrence, or any palpable or biopsy-detected local recurrence three years after radiation; any local recurrence within three years of RT if the most previous PSA was>2 ng/ml; and death from prostate cancer.
Time Frame: within 10 years following initiation of radiotherapy
Measure: Count of Participants; unit: Participants
Groups:
- Patients: All patients
Arm/Group | Patients
Number analyzed (Participants) | 2384
Participants | 315

2. Secondary Outcome: Number of Participants With Initiation of Salvage Therapy After Radiotherapy
Time Frame: within 10 years following initiation of radiotherapy
Measure: Count of Participants; unit: Participants
Groups:
- Patients: Eligible patients
Arm/Group | Patients
Number analyzed (Participants) | 2384
Participants | 267

3. Post Hoc Outcome: Prognostic Value of Hormone Therapy on the Risk of Clinical Failure.
Time Frame: within 10 years following initiation of radiotherapy
Measure: Number (95% Confidence Interval); unit: hazard ratio
Arm/Group | Patients
Number analyzed (Participants) | 2384
hazard ratio | 0.21 [0.14 to 0.30]
Statistical Analysis 1: Comparison: Patients; Test type: Other; Two-stage model. — Estimation was performed using a Bayesian approach. As such, p-values are not estimated; Hazard Ratio (HR) = 0.21, 95% CI 2-sided [0.14 to 0.30]; Two-stage model within a Bayesian framework to assess the role of the prostate-specific antigens profile on clinical failure while accounting for a secondary treatment prescribed by indication. Prostatespecific antigens modeled using a hierarchical piecewise linear trajectory with a random changepoint. Residual prostate-specific antigens variability was expressed as a function of prostate-specific antigens concentration. Covariates in the survival model included hormone therapy, baseline characteristics, and individual predictions of the prostate-specific antigens nadir and timing and prostate-specific antigens slopes before and after the nadir as provided by the longitudinal process

ADVERSE EVENTS:
Time Frame: up to 10 years following initiation of radiotherapy
Description: This study is a retrospective analysis focussing on the association between the longitudinal PSA trajectory and the time to clinical failure. As such, we did not report on safety.
  Serious and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Groups:
- All Patients: Eligible patients
Arm/Group | All Patients
All-Cause Mortality (participants affected / at risk) | 0/2384
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No